CLINICAL TRIAL: NCT01918072
Title: Controlled Trial of Tele-Support and Education for Womens Health Care in CBOCs
Acronym: WH CREATE P4
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CRE 12-031
Record Dates: First submitted 2013-07-16; First posted 2013-08-07 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Metrorrhagia; Urinary Incontinence; Remote Consultation; Videoconferencing; Women's Health; Menopause
Keywords: Women's Health; Hospitals, Veterans; Education; Remote consultation; Videoconferencing
MeSH Terms: conditions — Metrorrhagia; Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Not applicable - none
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Stepped wedge participants: Designated Women's Health Providers with one or more episodes of care for women patients during each period of the intervention.
  Designated Women's Health Provider: Primary care provider who are proficient in women's health, and should have a minimum of 10% of their patient panels being comprised by women.
  Interventions: Other: Clinical innovation
- Electronic consultation survey participants: Designated Women's Health Providers who completed surveys about use of electronic consultations.
  Designated Women's Health Provider: Primary care provider who are proficient in women's health, and should have a minimum of 10% of their patient panels being comprised by women.
  Interventions: Other: Clinical innovation
- Quality assessment participants: Primary care providers delivering women's health care for one or more of the following conditions: abnormal uterine bleeding; menopausal symptoms; urinary incontinence.
  Interventions: Other: Clinical innovation

INTERVENTIONS:
Other: Clinical innovation — Technology-based intervention that combines interactive communication with women's health specialists and ongoing education
  Other Names: "DWHP Support"

SUMMARY:
VA community-based outpatient clinics (CBOCs) typically serve only a small number of women Veterans, and generally do not have the women's health care resources that are available in larger settings. Women Veterans using these sites for primary care must sometimes travel to other sites to receive women's health care. That can create travel burdens, reduce continuity of care, and negatively affect patient outcomes. To address this, VA is implementing a clinical operations innovation that supports women's primary care providers with a technology-based intervention that combines interactive communication with women's health specialists and ongoing education. This research study is evaluating the implementation and effects of this women's healthcare delivery innovation. Findings from this research will inform VA women's health clinical practice and education, and will advance science in delivering technology-supported non-face-to-face care that is applicable to other clinical conditions and patient populations.

DETAILED DESCRIPTION:
Project Background/Rationale: Women Veterans are a rapidly growing proportion of VA patients. While entitled to receive care equivalent to their male counterparts, women Veterans may receive lower quality care, in part due to a VA primary care (PC) workforce that has limited experience caring for women, particularly their gender-specific conditions. This workforce may be especially challenged in community-based outpatient clinics (CBOCs), where access to women's health (WH) expertise may not be readily available. CBOC PC providers (PCPs) typically have small caseloads of women Veterans, making it difficult for these providers to maintain their WH knowledge and skills. To ensure quality care for women Veterans, VA mandated designated WH providers (DWHPs) in every VA facility, and instituted intensive training opportunities-"WH mini-residencies"-for these providers. Although highly valuable in delivering a standard level of specialized WH training, these one-time trainings are not sufficient, as knowledge attenuates over time. Serial education re-enforcement over time is needed to produce and maintain long-term gains in knowledge. Furthermore, additional supports, such as enhanced communication between PCPs and specialists, are necessary to achieve and sustain quality gains. To address these issues, VA is implementing a clinical operations innovation that is designed to improve CBOC-based DWHP delivery of comprehensive WH care. This innovation (entitled DWHP Support) combines: 1) advanced WH serial patient-based education that exposes DWHPs, over time, to a depth and breadth of WH cases and issues (SCAN-ECHO); and 2) interactive communication between CBOC DWHPs and VA Medical Center-based specialists for "just in time" support of DWHP WH care (electronic consultations). The intervention is technology-supported and delivered virtually. It is being implemented in a stepwise manner.

Objectives: Facilitators and barriers to use of DWHP Support, and its effect on patient management are unknown. The investigators hypothesize that DWHP Support will improve the quality and efficiency of WH care in CBOCs. The specific aims are:

Aim #1: To evaluate the effect of DWHP Support on WH care quality and efficiency, using a modified stepped wedge design; Aim #2: To explore the impact of DWHP Support in changing DWHP behavior and self-rated WH knowledge, skills, and self-efficacy; Aim #3: To assess attitudes about DWHP Support and its use, specialist time for its implementation, and other features that could influence DWHP Support's effectiveness, sustainability and spread; Aim #4: To develop tools to measure quality of WH care in VA.

Methods: The investigators will conduct an observational study of DWHP Support for CBOC DWHPs. The investigators will use a mixed methods analytic approach (combining a modified stepped wedge quantitative analysis with provider surveys and interviews) to measure the intervention's effect after 1 year, while also evaluating the implementation process and use of the intervention. The investigators will use quality assessment methods to translate existing evidence-based WH performance guidelines into quality measurement tools applicable to VA WH care.

Anticipated Impact: This proposal aims to evaluate an innovation to improve WH care in CBOCs that uses a technology-based educational and interactive communication intervention designed for WH providers. To measure the intervention's effectiveness, this project will develop WH quality measures that will be valuable tools for other VA efforts to improve WH care. The findings on effectiveness and implementation could influence VA's approach and use of technology-supported interventions for other clinical conditions and in other special populations.

ELIGIBILITY:
Inclusion Criteria:

US Department of Veterans Affairs Women's Health primary care provider in who participates in Veterans Affairs SCAN-ECHO learning sessions or uses Veterans Affairs gynecology electronic consults.

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VA Women's Health primary care provider in who participates in VA SCAN-ECHO learning sessions or uses VA gynecology electronic consults.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Washington, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordasco KM, Zuchowski JL, Hamilton AB, Kirsh S, Veet L, Saavedra JO, Altman L, Knapp H, Canning M, Washington DL. Early lessons learned in implementing a women's health educational and virtual consultation program in VA. Med Care. 2015 Apr;53(4 Suppl 1):S88-92. doi: 10.1097/MLR.0000000000000313. PMID 25767983
- [Result] deKleijn M, Lagro-Janssen AL, Canelo I, Yano EM. Creating a roadmap for delivering gender-sensitive comprehensive care for women Veterans: results of a national expert panel. Med Care. 2015 Apr;53(4 Suppl 1):S156-64. doi: 10.1097/MLR.0000000000000307. PMID 25767971
- [Result] Yano EM. A partnered research initiative to accelerate implementation of comprehensive care for women veterans: the VA women's health CREATE. Med Care. 2015 Apr;53(4 Suppl 1):S10-4. doi: 10.1097/MLR.0000000000000340. No abstract available. PMID 25767962
- [Result] Zuchowski JL, Hamilton AB, Washington DL, Gomez AG, Veet L, Cordasco KM. Drivers of Continuing Education Learning Preferences for Veterans Affairs Women's Health Primary Care Providers. J Contin Educ Health Prof. 2017 Summer;37(3):168-172. doi: 10.1097/CEH.0000000000000164. PMID 28817394
- [Result] Washington DL, Danz M, Jackson L, Cordasco KM. Development of Quality Indicators for the Care of Women with Abnormal Uterine Bleeding by Primary Care Providers in the Veterans Health Administration. Womens Health Issues. 2019 Mar-Apr;29(2):135-143. doi: 10.1016/j.whi.2018.11.002. Epub 2018 Dec 15. PMID 30563732
- [Result] Cordasco KM, Yuan AH, Danz MJ, Farmer MM, Jackson L, Yee EF, Washington DL. Guideline Adherence of Veterans Health Administration Primary Care for Abnormal Uterine Bleeding. Womens Health Issues. 2019 Mar-Apr;29(2):144-152. doi: 10.1016/j.whi.2018.12.004. Epub 2019 Feb 2. PMID 30723059
- [Result] Cordasco KM, Yuan AH, Danz MJ, Jackson L, Yee EF, Tcheung LS, Washington DL. Veterans Health Administration Primary Care Provider Adherence to Prescribing Guidelines for Systemic Hormone Therapy in Menopausal Women. J Healthc Qual. 2019 Mar/Apr;41(2):99-109. doi: 10.1097/JHQ.0000000000000183. PMID 30839493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers (PCPs) delivering women's health care from June 2013 - September 2015 in VA healthcare systems that implemented the DWHP Support women's health clinical innovation, which is a technology-based program that combines interactive communication with women's health specialist and ongoing education.
Pre-assignment Details: STEPPED WEDGE CONTROLLED TRIAL INCLUSION CRITERIA: Designated Women's Health Providers (DWHPs) with one or more episodes of care for women patients during each period of the intervention. ELECTRONIC CONSULTATION SURVEY INCLUSION CRITERIA: DWHPs who submitted and received a response to a gynecology electronic consult during the study timeframe.
Period: Controlled Trial Step One - Six Months
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 11 | 0 | 0
Intervention (First primary care provider group steps into intervention) | 1 | 0 | 0
Control | 10 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Controlled Trial Step Two - Six Months
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 11 | 0 | 0
Intervention (Second primary care provider group steps into intervention) | 7 | 0 | 0
Control | 4 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Controlled Trial Step Three - Six Months
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 11 | 0 | 0
Intervention (Third primary care provider group steps into intervention) | 9 | 0 | 0
Control | 2 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Controlled Trial Step Four - Six Months
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 11 | 0 | 0
Intervention (Fourth primary care provider group steps into intervention) | 11 | 0 | 0
Control | 0 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Controlled Trial Step Five - Four Months
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 11 | 0 | 0
Intervention (All primary care provider groups fully in intervention) | 11 | 0 | 0
Control | 0 | 0 | 0
Completed | 11 | 0 | 0
Not Completed | 0 | 0 | 0
Period: E-consult Assessment Period
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 0 | 42 | 0
Completed | 0 | 42 | 0
Not Completed | 0 | 0 | 0
Period: Quality Assessment Period
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
Started | 0 | 0 | 202
Completed | 0 | 0 | 202
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VA Primary Care Providers Delivering Women's Health Care: Primary care providers in VA healthcare systems that implemented the DWHP Support women's health clinical innovation (a technology-based program that combines interactive communication with women's health specialist and ongoing education).
Arm/Group | VA Primary Care Providers Delivering Women's Health Care
Number analyzed (Participants) | 202
Age, Customized [Count of Participants; unit: Participants] — Population: STEPPED WEDGE CONTROLLED TRIAL: DWHPs with one or more episodes of care for women patients during each period of the intervention.
  E-CONSULT SURVEY: DWHPs who completed surveys about e-consult use.
  QUALITY ASSESSMENT: PCPs delivering women's health care for abnormal uterine bleeding, menopausal symptoms, or urinary incontinence.
  Participants
    Stepped wedge: number analyzed (Participants) | 11
    Stepped wedge: <18 years | 0
    Stepped wedge: 18 years or older | 11
    Electronic consultations: number analyzed (Participants) | 42
    Electronic consultations: <18 years | 0
    Electronic consultations: 18 years or older | 42
    Quality assessment: <18 years | 0
    Quality assessment: 18 years or older | 202
Sex: Female, Male [Count of Participants; unit: Participants] — Population: STEPPED WEDGE CONTROLLED TRIAL: DWHPs with one or more episodes of care for women patients during each period of the intervention.
  QUALITY ASSESSMENT: PCPs delivering women's health care for abnormal uterine bleeding, menopausal symptoms, or urinary incontinence.
  E-CONSULT SURVEY: Sex data were not collected.
  Participants
    Stepped wedge: number analyzed (Participants) | 11
    Stepped wedge: Female | 10
    Stepped wedge: Male | 1
    Quality assessment: Female | 141
    Quality assessment: Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 202
Designated Women's Health Provider (DWHP) status [Count of Participants; unit: Participants] — Population: This baseline measure was assessed for participants in the stepped wedge controlled trial.
  Participants
    number analyzed (Participants) | 11
    DWHP | 11
    Non-DWHP | 0
Professional degree [Count of Participants; unit: Participants] — Population: This baseline measure was assessed for participants in the stepped wedge controlled trial.
  Participants
    number analyzed (Participants) | 11
    MD or DO | 4
    NP or PA | 7
Provider monthly encounters with women [Mean (Full Range); unit: months] — Population: This baseline measure was assessed for participants in the stepped wedge controlled trial.
  months
    number analyzed (Participants) | 11
    (all) | 159 [38 to 377]
Healthcare setting [Count of Participants; unit: Participants] — Population: This baseline measure was assessed for participants in the stepped wedge controlled trial.
  Participants
    number analyzed (Participants) | 11
    VA Medical Center | 7
    VA Community Based Outpatient Clinic | 4
Comprehensive women's health clinic setting [Count of Participants; unit: Participants] — Population: This baseline measure was assessed for participants in the stepped wedge controlled trial.
  Participants
    number analyzed (Participants) | 11
    VA comprehensive WH clinic | 5
    VA general primary care clinic | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Women's Health Care (Control Period vs. Intervention Period)
Description: Quality of care as defined by adherence to practice guidelines. This measure is the difference in the percent of applicable quality indicators for whom the guideline adherent action was performed by primary care providers at baseline versus after entering into the intervention.
Time Frame: Baseline through four months after the final time step when participants entered into the intervention (28 months)
Measure: Mean (Standard Error); unit: percent of care adherent to guidelines
Arm/Group | Stepped Wedge Participants
Number analyzed (Participants) | 11
percent of care adherent to guidelines | 7.1 (8.6)

2. Secondary Outcome: Change in Quality of Women's Health Care (Controlled Trial Steps)
Description: Quality of care as defined by adherence to practice guidelines. This measure is the difference in the percent of applicable quality indicators for whom the guideline adherent action was performed by primary care providers, with each subsequent step, over the course of the controlled trial.
Time Frame: Baseline through four months after the final time step when participants entered into the intervention (28 months)
Measure: Mean (Standard Error); unit: percent of care adherent to guidelines
Arm/Group | Stepped Wedge Participants
Number analyzed (Participants) | 11
percent of care adherent to guidelines | 9.6 (4.1)

3. Secondary Outcome: Provider Referral Behavior
Description: This measure is the number of providers that changed their referral plan for an in-person specialist-to-patient visit after an electronic consultation.
Time Frame: 1-7 days after receiving a response to the electronic consult
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Consultation Survey Participants
Number analyzed (Participants) | 42
Participants | 13

4. Secondary Outcome: Quality of Abnormal Uterine Bleeding Care
Description: Quality of abnormal uterine bleeding care as defined by adherence to practice guidelines. This measure is the mean percent of applicable quality indicators for whom the guideline adherent action was performed by primary care providers.
Time Frame: 28-month study timeframe
Population: The analysis included primary care providers providing care for abnormal uterine bleeding episodes during the 28-month study timeframe.
Measure: Mean (95% Confidence Interval); unit: percent of care adherent to guidelines
Groups:
- Quality Assessment Participants: Primary care providers delivering women's health care for abnormal uterine bleeding.
Arm/Group | Quality Assessment Participants
Number analyzed (Participants) | 74
percent of care adherent to guidelines | 53 [51 to 56]

5. Secondary Outcome: Quality of Menopausal Symptoms Care
Description: Quality of menopausal symptoms care as defined by adherence to practice guidelines. This measure is the mean percent of applicable quality indicators for whom the guideline adherent action was performed by primary care providers.
Time Frame: 28-month study timeframe
Population: The analysis included primary care providers providing care for menopausal symptoms episodes during the 28-month study timeframe.
Measure: Mean (95% Confidence Interval); unit: percent of care adherent to guidelines
Groups:
- Quality Assessment Participants: Primary care providers delivering women's health care for menopausal symptoms.
Arm/Group | Quality Assessment Participants
Number analyzed (Participants) | 81
percent of care adherent to guidelines | 58 [55 to 60]

6. Secondary Outcome: Quality of Urinary Incontinence Care
Description: Quality of urinary incontinence care as defined by adherence to practice guidelines. This measure is the mean percent of applicable quality indicators for whom the guideline adherent action was performed by primary care providers.
Time Frame: 28-month study timeframe
Population: The analysis included primary care providers providing care for urinary incontinence episodes during the 28-month study timeframe.
Measure: Mean (95% Confidence Interval); unit: percent of care adherent to guidelines
Groups:
- Quality Assessment Participants: Primary care providers delivering women's health care for urinary incontinence.
Arm/Group | Quality Assessment Participants
Number analyzed (Participants) | 68
percent of care adherent to guidelines | 39 [36 to 42]

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study. To indicate that adverse events were not collected as part of the study, "0" is entered for the total number of participants at risk and affected for the three arms/groups listed in all adverse events tables.
Arm/Group | Stepped Wedge Participants | Electronic Consultation Survey Participants | Quality Assessment Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT01918072/Prot_SAP_000.pdf